CLINICAL TRIAL: NCT04024579
Title: Prospective, Single-arm, Medical Device Investigation According to § 23b MPG [German Medical Devices Act] on Efficacy and Safety of Treatment of Actinic Keratosis With a 5% Potassium Hydroxide Solution (AKOHDerm)
Brief Title: Treatment of Actinic Keratosis With 5% KOH Solution
Acronym: TAKKOH
Status: Completed | Type: Observational
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Collaborators: Gesellschaft für Therapieforschung mbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TAKKOH
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective single-arm multicenter medical device study to investigate the clinical efficacy and safety of the treatment of actinic keratosis with a 5% potassium hydroxide solution.

In total, 68 patients with actinic keratosis grade I/II, who meet all inclusion criteria and do not meet none of the exclusion criteria are to be enrolled and topically treated twice daily for up to 3 cycles of 14 days of treatment followed by 14 non-treatment days.

The primary objective is treatment success at the individual end-of-treatment visit of all AK lesions present at baseline and treated with the investigational product.

Beside this, adverse events will be collected at each visit and evaluated in order to investigate clinical safety.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age: 30 to 80 years
* Adults with AK grade I (mild) or II (moderate)

Exclusion Criteria:

* Number of lesions requiring treatment > 10
* Lesion to be treated > 20 mm (maximum diameter)
* Lesions directly adjoining to the eyes, eyelids, nostrils, mouth or mucosal tissue,
* Need for topical treatment of a cancerous area
* Presence of a relapsing, persistent, indurated, thickened, painful, bleeding, ulcerated and/or rapidly growing lesion
* Presence of a persistent or relapsing lesion despite appropriate treatment with AKOHDerm or another appropriate treatment
* High risk of progression of AK according as assessed by a medical doctor
* Pharmacological or physical local therapy of AK in the area foreseen for treatment dur-ing the last 12 weeks
* Treatment with systemic corticosteroids during the last 2 weeks
* Planned concomitant treatment of the same AK lesions during the study in addition to study treatment
* Other skin diseases in the area of application which might interfere with clinical signs
* Known predisposition for hypertrophic scarring / keloidosis
* Primary or secondary immunodeficiency
* Treatment with interferons, interferon inducers or immunomodulators during the last 4 weeks
* Pregnancy and lactation
* No reliable contraception in women of child-bearing potential
* Other serious diseases which are according to the investigator in conflict with the par-ticipation
* Obvious unreliability or lack of cooperation - known addiction to alcohol, medicinal products or drugs
* Dependent relationship with sponsor or investigator
* Participation in a clinical trial within the last 30 days
* Previous participation in this study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of the participating study sites (medical practice and experienced in the management and treatment of patients suffering from the disease as mentioned in the inclusion criterion), who fulfill all inclusion criteria and do not fulfill any of the exclusion criteria, are eligible for participation in the TAKKOH study
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-08-25 (Actual)

PRIMARY OUTCOMES:
Efficacy (Patients with treatment success): defined as dermatoscopically confirmed complete remission of all AK lesions by the investigator | Visit 14 days after EOT (End of treatment); up to 12 weeks depending treatment cycles nessesary
  Treatment success (yes, no) at the individual end-of-treatment visit (VE), defined as dermatoscopically confirmed complete remission of all AK lesions by the investigator, which were present at V0 and treated with the investigational product (complete clearance).

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich Abeck, Prof., Principal Investigator — Professor of dermatology and allergology
Locations (6):
- Germany (6):
  - Dermatologisches Zentrum, Bonn
  - Hautzentrum Dülmen, Dülmen
  - Hautärztliche Praxis, Friedrichshafen
  - Hautzentrum Nymphenburg, München
  - Haut- und Laserzentrum Potsdam, Potsdam
  - Hautarzt-Praxis, Stuttgart